CLINICAL TRIAL: NCT06428617
Title: A Multi-site, Prospective Registry of Patients Undergoing Gastric Fundal Mucosal Ablation at True You Weight Loss
Brief Title: Fundus Ablation Registry (Gastric Fundus Mucosal Ablation for Weight Loss)
Status: Recruiting | Type: Observational
Sponsor: True You Weight Loss (Other)
Responsible Party: Sponsor
Other Study IDs: RGT-002
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-05

CONDITIONS: Obesity
Keywords: obesity; ghrelin; hunger; ablation; True You Weight Loss; hunger hormone; fundus; fundus ablation; fundic ablation; GFMA
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to construct a multi-site, prospective registry to evaluate the clinical outcomes of patients who have undergone gastric fundus mucosal ablation at True You Weight Loss.

DETAILED DESCRIPTION:
Obesity is a chronic, progressive, multifactorial disease that contributes to increasing morbidity, mortality, and economic costs worldwide. The oxyntic mucosa of the gastric fundus is the principal site for the production of the orexigenic peptide hormone ghrelin. Ghrelin activates hunger-promoting pathways of the hypothalamus and opposes the satiety-promoting actions of other gastrointestinal peptides, leading to calorie-ingesting behaviors and weight gain. A method to reduce ghrelin production and decrease fundal compliance and capacity through mucosal devitalization may confer benefit to patients seeking treatment for obesity. This is a multi-site, prospective registry of patients who have elected to undergo Gastric Fundus Mucosal Ablation (GFMA) at a True You Weight Loss site in Cary, NC or Atlanta, GA. Study participants will consist of up to 200 adult patients of ages 18 to 65 years old who have elected to undergo GFMA at a True You Weight Loss site (Cary, NC or Atlanta, GA) prior to their involvement in the study. Participants that meet the criteria below will be deemed eligible for participation after consultation with the study investigator. Study participants will receive follow-up care according to standard of care practices, regardless of their involvement in the research study. Standard of care nutritional practice includes a comprehensive lifestyle program with long-term nutritional support and monitoring. Patient weights and adverse events will be collected at each visit. Adverse events will be communicated to medical team members in between dedicated visits. We aim to establish a multi-site, prospective registry to longitudinally describe GMFA in adults with obesity, including patient characteristics, weight loss, improvement in weight-related medical conditions, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 65 years old
2. BMI ≥ 27 and ≤55 kg/m²
3. Willingness to comply with the substantial lifelong dietary restrictions required by the procedure.
4. Ability to give informed consent
5. Women of childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods.
6. Those who plan to receive the gastric fundus mucosal ablation procedure at True You Weight Loss regardless of the research

Exclusion Criteria:

1. Patients that do not meet eligibility requirements for the study as per the Principal Investigator's standard selection criteria
2. Active psychological issues preventing participation in a life-style modification program as determined by a psychologist.
3. Patients who are pregnant or breast-feeding.
4. Eating disorders including night eating syndrome (NES), bulimia, binge eating disorder, or compulsive overeating.
5. Patients with previous or current tobacco use
6. Patients with prior gastric surgery (e.g., vertical sleeve gastrectomy, gastric bypass, hiatal hernia repair, Nissen fundoplication, adjustable gastric band).
7. Patients on therapeutic anticoagulation or antithrombotics that cannot be interrupted for at least 12 weeks following GFMA.
8. Patients who cannot commit to 12 weeks of post-GMFA pharmacologic ulcer prophylaxis
9. At the discretion of the PI for subject safety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will consist of up to 200 adult patients of ages 18 to 65 years old who have elected to undergo Gastric Fundus Mucosal Ablation (GFMA) at a True You Weight Loss site (Cary, NC or Atlanta, GA) prior to their involvement in the study. Participants that meet the criteria below will be deemed eligible for participation after consultation with the study investigator. All eligibility criteria must be met at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Total Body Weight Loss (TBWL) from Baseline | 12 Months
  Measured percent change in total body weight over time following Gastric Fundus Mucosal Ablation. %TBWL = (pre-op weight - post op body weight) / (pre-op weight) * 100 measured as a percentage.

SECONDARY OUTCOMES:
Percent Change in Total Body Weight Loss (TBWL) from Baseline | 3 Months, 6 Months, 9 Months, 12 Months, 15 Months, 24 Months
  Measured percent change in total body weight over time following Gastric Fundus Mucosal Ablation. %TBWL = (pre-op weight - post op body weight) / (pre-op weight) * 100 measured as a percentage.
Percent Excess Weight Loss from Baseline (EWL) | 3 Months, 6 Months, 9 Months, 12 Months, 15 Months, 24 Months
  Measured excess weight loss percentage from baseline following Gastric Fundic Mucosal Ablation. %EWL = (pre-op weight - post op body weight) / (pre-op weight - ideal body weight) * 100
  Ideal Body Weight (IBW):
  Males: IBW = 50 kg + 2.3 kg for each inch over 5 feet Females: IBW = 45.5 kg + 2.3 kg for each inch over 5 feet
Change in Body Mass Index (BMI) from Baseline | 3 Months, 6 Months, 9 Months, 12 Months, 15 Months, 24 Months
  Measured Body Mass Index (BMI) from baseline following Gastric Fundic Mucosal Ablation. Body Mass Index (BMI) = (Weight in kilograms) / ((Height in meters)^2)

CONTACTS AND LOCATIONS:
Locations (1):
- True You Weight Loss, Cary, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No